CLINICAL TRIAL: NCT01982591
Title: Assessing Heavy Metal Contributions to Neurotoxicity in Breast Cancer Patients Undergoing Adjuvant or Neoadjuvant Chemotherapy
Brief Title: Heavy Metal Exposure in Predicting Peripheral Neuropathy in Patients With Stage I-III Breast Cancer Undergoing Chemotherapy
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ERP-BR-059; NCI-2013-01957 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB#10-039; BR-059; ERP-BR-059 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2013-10-24; First posted 2013-11-13 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Male Breast Cancer; Neurotoxicity; Peripheral Neuropathy; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Neurotoxicity Syndromes; Peripheral Nervous System Diseases; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (heavy metal and neurotoxicity): Patients undergo serum and urine sample collection for heavy metal analysis by ICP-MS at baseline and at the completion of treatment. Patients also complete neurotoxicity assessment questionnaire at baseline and at the completion of treatment.
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This research trial studies heavy metal exposure in predicting peripheral neuropathy in patients with stage I-III breast cancer undergoing chemotherapy. Studying samples of blood and urine in the laboratory for heavy metal exposure from patients receiving chemotherapy may help doctors find out whether side effects from chemotherapy are related to heavy metal exposure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the correlation, if any, of specific heavy metals with high grade symptoms of peripheral neuropathy, defined as grade >= 3 peripheral neuropathy, (utilizing the Common Terminology Criterial for Adverse Events [CTCAE] version [v.] 4.0) in a cohort of breast cancer patients undergoing (neo)adjuvant taxane chemotherapy.

SECONDARY OBJECTIVES:

I. To characterize the range of specific heavy metals in a cohort of breast cancer patients undergoing (neo)adjuvant chemotherapy treatment.

II. To evaluate the reproducibility of sera and urine testing of heavy metal levels by inductively coupled plasma mass spectrometry (ICP-MS) testing in a cohort of breast cancer patients undergoing (neo)adjuvant taxane chemotherapy.

OUTLINE:

Patients undergo serum and urine sample collection for heavy metal analysis by ICP-MS at baseline and at the completion of treatment. Patients also complete neurotoxicity assessment questionnaire at baseline and at the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed invasive mammary carcinoma; any histologic sub-type allowed
* Patients must be diagnosed with stage I, II or III breast cancer
* Patients must be undergoing treatment with an adjuvant or neoadjuvant cytotoxic chemotherapy that includes a taxane, specifically paclitaxel, nab-paclitaxel (Abraxane), or docetaxel
* Patients may have received prior endocrine and/or radiation therapy
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have been previously treated with cytotoxic chemotherapy
* Patients with pre-existing peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2011-01-03 (Actual); Primary Completion 2015-03-24 (Actual); Study Completion 2015-03-24 (Actual)

PRIMARY OUTCOMES:
Level of heavy metal in blood and urine | The levels will be measured on a blood and urine sample obtained on the first day of chemotherapy, which is considered the first day of the study. The actual laboratory processing of the samples will occur in batches throughout the duration of the study.
  Heavy metal levels will be characterized in participants being treated at participating sites. Means and variances and ranges of these levels will be tabulated.
Incidence of high grade neurotoxicity, defined as grade >= 3 peripheral neuropathy, graded according to CTCAE v. 4.0 | Last day of chemotherapy approx.4-6 months from initiation, depending on chemotherapy regimen. Neurotoxicity grade will be assessed intermittently during course of therapy, with note of maximum grade made by clinician.
  Neurotoxicity grade during chemotherapy will be obtained from the medical record and study doctor's notes. The maximum grade during the course of chemotherapy will be recorded. Frequencies of toxicities will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Goldstein, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania